CLINICAL TRIAL: NCT01927913
Title: A 48-week, Open-label, 2-arm, Parallel-group, Randomized Exploratory Study to Assess Liver Iron Concentration Measured by FerriScan® (R2) Magnetic Resonance Imaging in B-thalassemia Subjects Administered SPD602 (SSP-004184AQ) or Exjade® (Deferasirox) for Treatment of Chronic Transfusional Iron Overload
Brief Title: Treatment of Iron Overload Requiring Chelation Therapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was withdrawn until the evaluation of the nonclinical rat findings is complete.
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPD602-204; FBS0701 (SSP-004184); 2013-000743-33 (EudraCT Number)
Record Dates: First submitted 2013-08-20; First posted 2013-08-23 (Estimated); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Transfusional Iron Overload; Iron Overload; Iron Chelation; Beta-thalassemia; Transfusional Hemosiderosis; Iron Metabolism Disorders; Metabolic Diseases
MeSH Terms: conditions — Iron Overload; beta-Thalassemia; Iron Metabolism Disorders; Metabolic Diseases | interventions — Deferasirox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SPD602 (Experimental)
  Interventions: Drug: SPD602
- Deferasirox (Active Comparator)
  Interventions: Drug: Deferasirox

INTERVENTIONS:
Drug: SPD602 — 32, 50 or 75 mg/kg/day BID, capsule
  Other Names: SSP-004184AQ
  Arms: SPD602
Drug: Deferasirox — Per approved country specific label
  Other Names: Exjade®
  Arms: Deferasirox

SUMMARY:
The purpose of this open-label study is to assess liver iron concentration using MRI imaging in subjects with beta-thalassemia when administered with either SPD602 or deferasirox for the treatment of chronic transfusional iron overload.

ELIGIBILITY:
Inclusion Criteria:

These criteria are to be met at the Screening Visit (Visit 1), the Washout Visit (Visit 2), and the Baseline Visit (Visit 3), if reassessed.

* An understanding, ability, and willingness to fully comply with study procedures and restrictions.
* Ability to voluntarily provide written, signed, and dated (personally or via a legally authorized representative) informed consent as applicable to participate in the study before completing any study-related procedures.
* Subjects 18 years of age or older at the time of signing consent.
* Female subjects should be one of the following:

  1. Post-menopausal (12 consecutive months of spontaneous amenorrhea)
  2. Surgically sterile, or
  3. Females of child-bearing potential must have a negative serum Beta-HCG pregnancy test at the Screening Visit (Visit 1) and a negative urine pregnancy test at the Baseline Visit (Visit 3). Females of child-bearing potential must agree to abstain from sexual activity that could result in pregnancy or agree to use acceptable methods of contraception.
* Subjects with beta-thalassemia who have received at least 100mL/kg of packed red blood cells (or >20 transfusion units) and who have iron overload (transfusional hemosiderosis) requiring chronic treatment with an iron chelator.
* Serum ferritin >500µg/L at the Screening Visit (Visit 1).
* Baseline LIC (last MRI assessment prior to Day 1) greater than or equal to 2.0mg and less than 30.0mg iron per g (equivalent dry weight, liver) determined by FerriScan® R2 MRI.

  8. Mean of the previous 3 pre-transfusion hemoglobin concentrations greater than or equal to 7.5g/dL assessed at the Screening Visit (Visit 1) (1 value from clinical laboratory tests taken at the Screening Visit [Visit 1] and the previous 2 historical values available).

Exclusion Criteria:

* Severe iron overload including: (a) cardiac T2* MRI less than 10.0ms; or (b) LIC by FerriScan® R2 MRI greater than or equal to 30.0mg/g liver (dw) as assessed at the Screening Visit (Visit 1).
* Iron overload from causes other than transfusional siderosis.
* Subjects with thalassemia intermedia
* Unable to undergo MRI assessment.
* Cardiac LVEF less than 50% at baseline testing by MRI.
* Subjects with documented liver failure (presence of portal hypertension, hepatic edema, ascites, cirrhosis), Child-Pugh C hepatic impairment, or biliary disorder.
* Platelet count <100 x 109/L at the Screening Visit (Visit 1).
* Absolute neutrophils counts of <1500mm3 at the Screening Visit (Visit 1).
* Evidence of renal insufficiency eg, creatinine clearance <60mL/min or serum creatinine >1.5x ULN at the Screening Visit (Visit 1).
* Clinically significant laboratory assessments at the Screening Visit (Visit 1).
* Significant proteinuria: urinary protein/creatinine ratio >1.0 in a non-first void urine sample at the Screening Visit (Visit 1).
* Current or recurrent disease that could affect the action, absorption, or disposition of the investigational product, or clinical or laboratory assessments.
* Current or relevant history of physical or psychiatric illness, any medical disorder that may require treatment or make the subject unlikely to fully complete the study, or any condition, including pregnancy, that presents undue risk from the investigational product or procedures.
* Current use of any medication contraindicated in the deferasirox prescribing information/SmPC.
* Known or suspected intolerance or hypersensitivity to SSP-004184AQ, deferasirox, closely-related compounds, or any of the stated ingredients in either medication.
* Known history of alcohol or other substance abuse within the last year.
* Within 30 days prior to the Baseline Visit (Visit 3):

  1. Have used an investigational product
  2. Have been enrolled in a clinical study (including vaccine studies) that, in the investigator's opinion, may impact this study.
* History of malignancy within the past 5 years, with the exception of basal cell or squamous cell skin carcinoma or cervical carcinoma in situ or completely resected colon carcinoma in situ.
* Insufficient venous access that precludes prescribed blood draws for safety laboratory assessments.
* Pregnant or lactating females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-11-20 (Estimated); Primary Completion 2015-10-30 (Estimated); Study Completion 2015-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in Liver Iron Concentration (LIC) from Baseline Utilizing R2 Magnetic Resonance Imaging (MRI) | 48 Weeks

SECONDARY OUTCOMES:
Response Rate Utilizing R2* MRI | 48 weeks
Change in Cardiac Iron Concentration (CIC) from baseline Utilizing T2* MRI | 48 weeks
Change in Serum Ferritin Levels from Baseline | 48 weeks
Change in Pancreas Iron Concentration (PIC) from Baseline Utilizing R2* MRI | 48 weeks
Left Ventricular Ejection Fraction (LVEF) Utilizing MRI | 48 weeks
Gastrointestinal Symptom Rating Scale | 48 weeks
Total Neuropathy Score nurse (TNSn) | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda

REFERENCES:
- [Derived] Padhani ZA, Gangwani MK, Sadaf A, Hasan B, Colan S, Alvi N, Das JK. Calcium channel blockers for preventing cardiomyopathy due to iron overload in people with transfusion-dependent beta thalassaemia. Cochrane Database Syst Rev. 2023 Nov 17;11(11):CD011626. doi: 10.1002/14651858.CD011626.pub3. PMID 37975597